CLINICAL TRIAL: NCT03132662
Title: Comparative Trial of Omega-3 Polyunsaturated Fatty Acids vs a Very Low Calorie Liquid Diet for Liver Volume Reduction Prior to Bariatric Surgery
Brief Title: Omega-3 vs Very Low Calorie Diet for Liver Size Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Collaborators: Neptune (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJHH_2042
Record Dates: First submitted 2017-04-03; First posted 2017-04-28 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2017-04

CONDITIONS: Obesity, Morbid; Obesity; NAFLD; NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Obesity, Morbid; Obesity; Non-alcoholic Fatty Liver Disease | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Very Low Calorie Diet (Active Comparator): The first group will continue according to the standard bariatric preoperative protocol and will be assigned a VLCLD of 900 cal/day (Optifast ® 4 servings/day each containing: 225 cal + 0.35 g linolenic acid) for 2-3 weeks prior to surgery according to the surgeon's preferences.
  Interventions: Dietary Supplement: Very Low Calorie Diet
- Omega-3 (Experimental): The second group will be assigned to 3 gr. daily oral intake of Ω-3 PUFAs ((Oceano3 ® 1000 mg Krill Oil tabs (150 mg EPA + 90 mg DHA) 3 times a day) for 4 weeks with only regular dietary suggestions before surgery.
  Interventions: Dietary Supplement: Omega-3
- No-treatment (No Intervention): The third group will not receive treatment for liver size reduction prior to surgery.

INTERVENTIONS:
Dietary Supplement: Omega-3 — 3 gr/day of Omega-3
  Arms: Omega-3
Dietary Supplement: Very Low Calorie Diet — 4 servings/day Optifast
  Arms: Very Low Calorie Diet

SUMMARY:
A recent review demonstrated that Non-alcoholic fatty liver disease (NAFLD) affects 10-35% of the adult population worldwide, with the prevalence approaching 85-100% in obese populations. Current standard treatment for liver reduction before surgery is the use of a very low calorie liquid diet (VLCLD). Multiple studies have shown that a 2-4 week diet with a VLCD will reduce liver volume, in preparation for surgery. Omega-3 (Ω-3) polyunsaturated fatty acids (PUFAs) have been suggested as a treatment for NAFLD. The primary aim of this study is to compare Ω-3 PUFAs and a VLCLD and their effect on left lobe live size before bariatric surgery.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is defined by the pathological accumulation of fat in the liver when no other explanatory disease is present: it encompasses isolated hepatic steatosis, non-alcoholic steatohepatitis (NASH) cirrhosis, and is a frequent accompaniment of obesity and insulin resistance. A recent review demonstrated that NAFLD affects 10-35% of the adult population worldwide, with the prevalence approaching 85-100% in obese populations.

Although frequently asymptomatic and relatively benign, NAFLD has the potential to progress to cirrhosis. Cirrhosis, when decompensated, has a poor prognosis.

Also, NAFDL will be accompanied invariably with increased liver volume, which will directly increase the level of difficulty of upper gastrointestinal surgery, such as bariatric surgery, specifically for the visualization of the gastro-esophageal junction. Bleeding is also more frequent with larger fattier left liver lobes. The combination of these factors may lead to conversion to open surgery, thus: increasing postoperative pain due to larger incisions, prolonging postoperative recovery times and increasing the risks of infection and hernias.

Current standard treatment for liver reduction before surgery is the use of a very low calorie liquid diet (VLCLD). Multiple studies have shown that a 2-4 week diet with Optifast® will reduce liver volume, in preparation for surgery.

Omega-3 (Ω-3) polyunsaturated fatty acids (PUFAs) have been suggested as a treatment for NAFLD. They have several potential mechanisms of action, the most important being to alter hepatic gene expression, thereby switching intracellular metabolism from lipogenesis and storage to fatty acid oxidation and catabolism. There is also evidence that they improve insulin sensitivity, are anti-inflammatory and reduce TNF levels lipogenesis thus offering several potential therapeutic mechanisms.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet ALL of the following inclusion criteria:

* Fulfilled criteria for bariatric surgery as coined by National Institutes of Health conference (a body mass index (BMI) of 40 or more, OR a BMI of 35 or more with a serious health problem linked to obesity, such as type 2 diabetes, heart disease, or sleep apnea)
* Their age is ≥18 years and ≤70 years
* Able and willing to give written consent
* The patient is willing to perform the pre-operative tests required for this study.

Exclusion Criteria:

Participants who meet any of the following criteria at the time of the baseline visit are NOT eligible to be enrolled in this study:

* Prior bariatric surgery
* Patient must not have any acute or chronic alteration of liver function (i.e. cirrhosis, active or chronic hepatitis, congenital hepatic disease, etc.)
* Prior hepatic surgery
* Contra-indication to general anesthesia
* Any medical condition, which in the judgement of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure
* Pregnant or lactating female (Women of child bearing potential must take a pregnancy test prior to surgery)
* Patients receiving medication that would alter hepatic function significantly.
* Patients with ascites.
* History of alcohol abuse: >3 standard drinks/day in men or >2 standard drinks/day in women (one standard drink being defined as 12 ounces of 5% beer, 5 ounces of 12% wine or 1.5 ounces of 40% liquor).
* Patients consuming Ω-3 supplements on a regular basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Left liver lobe size | First ultrasound will be done before treatment. Second ultrasound will be done after the treatment period of 3 weeks, before bariatric surgery is completed
  Size measured by sonography in centimetres.

SECONDARY OUTCOMES:
NAFLD | First ultrasound will be done before treatment. Second ultrasound will be done after the treatment period of 3 weeks, before bariatric surgery is completed
  Liver density measures of sonography
Costs | After the treatment period of 3 weeks, before bariatric surgery is completed
  Amount paid out of pocket by patient for treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hong, MD, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellentani S, Marino M. Epidemiology and natural history of non-alcoholic fatty liver disease (NAFLD). Ann Hepatol. 2009;8 Suppl 1:S4-8. PMID 19381118
- [Background] Hui JM, Kench JG, Chitturi S, Sud A, Farrell GC, Byth K, Hall P, Khan M, George J. Long-term outcomes of cirrhosis in nonalcoholic steatohepatitis compared with hepatitis C. Hepatology. 2003 Aug;38(2):420-7. doi: 10.1053/jhep.2003.50320. PMID 12883486
- [Background] Masterton GS, Plevris JN, Hayes PC. Review article: omega-3 fatty acids - a promising novel therapy for non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2010 Apr;31(7):679-92. doi: 10.1111/j.1365-2036.2010.04230.x. PMID 20415840
- [Background] Parker HM, Johnson NA, Burdon CA, Cohn JS, O'Connor HT, George J. Omega-3 supplementation and non-alcoholic fatty liver disease: a systematic review and meta-analysis. J Hepatol. 2012 Apr;56(4):944-51. doi: 10.1016/j.jhep.2011.08.018. Epub 2011 Oct 21. PMID 22023985
- [Background] Clarke SD. Nonalcoholic steatosis and steatohepatitis. I. Molecular mechanism for polyunsaturated fatty acid regulation of gene transcription. Am J Physiol Gastrointest Liver Physiol. 2001 Oct;281(4):G865-9. doi: 10.1152/ajpgi.2001.281.4.G865. PMID 11557505
- [Background] Svegliati-Baroni G, Candelaresi C, Saccomanno S, Ferretti G, Bachetti T, Marzioni M, De Minicis S, Nobili L, Salzano R, Omenetti A, Pacetti D, Sigmund S, Benedetti A, Casini A. A model of insulin resistance and nonalcoholic steatohepatitis in rats: role of peroxisome proliferator-activated receptor-alpha and n-3 polyunsaturated fatty acid treatment on liver injury. Am J Pathol. 2006 Sep;169(3):846-60. doi: 10.2353/ajpath.2006.050953. PMID 16936261
- [Background] Bellentani S, Saccoccio G, Masutti F, Croce LS, Brandi G, Sasso F, Cristanini G, Tiribelli C. Prevalence of and risk factors for hepatic steatosis in Northern Italy. Ann Intern Med. 2000 Jan 18;132(2):112-7. doi: 10.7326/0003-4819-132-2-200001180-00004. PMID 10644271
- [Background] Lewis MC, Phillips ML, Slavotinek JP, Kow L, Thompson CH, Toouli J. Change in liver size and fat content after treatment with Optifast very low calorie diet. Obes Surg. 2006 Jun;16(6):697-701. doi: 10.1381/096089206777346682. PMID 16756727
- [Background] Colles SL, Dixon JB, Marks P, Strauss BJ, O'Brien PE. Preoperative weight loss with a very-low-energy diet: quantitation of changes in liver and abdominal fat by serial imaging. Am J Clin Nutr. 2006 Aug;84(2):304-11. doi: 10.1093/ajcn/84.1.304. PMID 16895876
- [Background] Cohen JC, Horton JD, Hobbs HH. Human fatty liver disease: old questions and new insights. Science. 2011 Jun 24;332(6037):1519-23. doi: 10.1126/science.1204265. PMID 21700865
- [Background] Capanni M, Calella F, Biagini MR, Genise S, Raimondi L, Bedogni G, Svegliati-Baroni G, Sofi F, Milani S, Abbate R, Surrenti C, Casini A. Prolonged n-3 polyunsaturated fatty acid supplementation ameliorates hepatic steatosis in patients with non-alcoholic fatty liver disease: a pilot study. Aliment Pharmacol Ther. 2006 Apr 15;23(8):1143-51. doi: 10.1111/j.1365-2036.2006.02885.x. PMID 16611275
- [Background] Spadaro L, Magliocco O, Spampinato D, Piro S, Oliveri C, Alagona C, Papa G, Rabuazzo AM, Purrello F. Effects of n-3 polyunsaturated fatty acids in subjects with nonalcoholic fatty liver disease. Dig Liver Dis. 2008 Mar;40(3):194-9. doi: 10.1016/j.dld.2007.10.003. Epub 2007 Dec 4. PMID 18054848
- [Background] Iannelli A, Martini F, Schneck AS, Ghavami B, Baudin G, Anty R, Gugenheim J. Preoperative 4-week supplementation with omega-3 polyunsaturated fatty acids reduces liver volume and facilitates bariatric surgery in morbidly obese patients. Obes Surg. 2013 Nov;23(11):1761-5. doi: 10.1007/s11695-013-0942-y. PMID 23686653